CLINICAL TRIAL: NCT01339299
Title: The Endocrine Efficacy of Either Recombinant Luteinizing Hormone (r-LH) or Low Dose Recombinant Human Chorionic Gonadotropin (r-hCG) Supplementation for Recombinant Follicle Stimulating Hormone (r-FSH) Stimulation in Normogonadotrophic Women Undergoing in Vitro Fertilization (IVF)/Intracytoplasmic Sperm Injection (ICSI) Therapy Following a Long-term Gonadotropin Releasing Hormone (GnRH) Agonist Down Regulation Protocol
Brief Title: Study to Examine Effect of Recombinant Luteinizing Hormone (r-Lh) and Recombinant Human Chorionic Gonadotropin (r-hCG) for Ovarian Stimulation in Assisted Reproduction Techniques (ART)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Peter Humaidan, Prof. M.D. D.M.Sc., Regionshospitalet Viborg, Skive
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 700642-603; 2009-009375-35 (EudraCT Number)
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2011-04

CONDITIONS: Controlled Ovarian Stimulation; Infertility
Keywords: COS; ART; Infertility
MeSH Terms: conditions — Infertility | interventions — Luteinizing Hormone; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- recombinant luteinizing hormone (Experimental): 150 IU r-LH, recombinant luteinising hormone, from treatment day 1 (stimulation day 1) until day of r-hCG administration (normally treatment day 10 to 14)
  Interventions: Drug: recombinant luteinizing hormone (r-LH)
- recombinant human chorionic gonadotrofin (Active Comparator): 25 IU of r-hCG from treatment day 1 (stimulation day 1) until day of r-hCG administration (normally treatment day 10 to 14 )
  Interventions: Drug: recombinant human chorionic gonadotropin (r-hCG)

INTERVENTIONS:
Drug: recombinant luteinizing hormone (r-LH) — administration of r-LH 150 IU/day subcutaneously , from S1 to r-hCG administration day (treatment day 10 to 14)
  Arms: recombinant luteinizing hormone
Drug: recombinant human chorionic gonadotropin (r-hCG) — administration of r-hCG 25 IU/day subcutaneously , from S1 to r-hCG administration day (treatment day 10 to 14)
  Arms: recombinant human chorionic gonadotrofin

SUMMARY:
The study is a prospective, randomised, controlled, and non-blinded multi-center pilot study to evaluate endocrine efficacy of recombinant luteinizing hormone versus recombinant human chorionic gonadotropin administered during controlled ovarian stimulation for IVF/ICSI in normogonadotrophic women.

ELIGIBILITY:
Inclusion Criteria:

* Women who plan to undergo IVF or ICSI treatment
* Woman's age > 18 years but ≤ 35 years
* Regular menstrual cycle (25-34 days)
* BMI 18 to 30 inclusive
* Signed patient information and informed consent forms

Exclusion Criteria:

* PCOS
* More than 2 prior IVF/ICSI attempts
* Diabetes mellitus, epilepsy, lever-, kidney-, heart- and metabolism disorders, according to the Investigator's assessment.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic Skive regional Hospital, Skive, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Recombinant Human Chorionic Gonadotrofin: 25 IU of r-hCG from treatment day 1 (stimulation day 1) until day of r-hCG administration (normally treatment day 10 to 14 )
  recombinant human chorionic gonadotropin (r-hCG) : administration of r-hCG 25 IU/day subcutaneously , from S1 to r-hCG administration day (treatment day 10 to 14)
- Recombinant Luteinizing Hormone: 150 IU r-LH, recombinant luteinising hormone, from treatment day 1 (stimulation day 1) until day of r-hCG administration (normally treatment day 10 to 14)
  recombinant luteinizing hormone (r-LH) : administration of r-LH 150 IU/day subcutaneously , from S1 to r-hCG administration day (treatment day 10 to 14)
Period: Overall Study
Arm/Group | Recombinant Human Chorionic Gonadotrofin | Recombinant Luteinizing Hormone
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombinant Human Chorionic Gonadotrofin | Recombinant Luteinizing Hormone | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.7 (3.1) | 30.1 (3.2) | 29.9 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: The Oestradiol Concentration on the Day of Ovulation Induction
Time Frame: treatment day 10 to 14
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Recombinant Human Chorionic Gonadotrofin | Recombinant Luteinizing Hormone
Number analyzed (Participants) | 50 | 50
pmol/L | 11482 (8210) | 12262 (8100)

ADVERSE EVENTS:
Arm/Group | Recombinant Human Chorionic Gonadotrofin | Recombinant Luteinizing Hormone
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes